CLINICAL TRIAL: NCT01153256
Title: The Influence of Magnesium Sulphate Pretreatment on Intubating Conditions During Rapid Sequence Induction
Brief Title: Intubating Condition After Magnesium Pre-treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: Mg_rocu
Record Dates: First submitted 2010-04-09; First posted 2010-06-30 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Easy of Laryngoscopy Manipulation; Vocal Cord Position or Movement; Patient Reaction to Intubation and Cuff Inflation; Mean Arterial Pressure; Heart Rate
MeSH Terms: interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- group M (Experimental)
  Interventions: Drug: magnesium sulphate
- Group R-0.6 (Placebo Comparator)
  Interventions: Drug: normal saline
- Group R-0.9 (Placebo Comparator)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: magnesium sulphate — The patients of group M receive 50 mg/kg of magnesium sulphate in 100 ml of isotonic saline over 10 min immediately before anaesthesia induction. After induction of anesthesia with alfentanil (10 μg/kg) and propofol (2 mg/kg), rocuronium 0.6 mg/kg is given over 5 s in a running infusion.
  Arms: group M
Drug: normal saline — Patients in the group R-0.6 receive the same volume of isotonic saline over the same period, and rocuronium 0.6 mg/kg is given after the induction of anesthesia with alfentanil (10 μg/kg) and propofol (2 mg/kg).
  Arms: Group R-0.6
Drug: normal saline — Patients in the group R-0.6 receive the same volume of isotonic saline over the same period, and rocuronium 0.9 mg/kg is given after the induction of anesthesia with alfentanil (10 μg/kg) and propofol (2 mg/kg).
  Arms: Group R-0.9

SUMMARY:
Magnesium had an inhibitory effect on neuromuscular transmission and caused a decrease in muscle fiber membrane excitability. It reduces the amount of acetylcholine that is released at the motor nerve terminal by decreasing the calcium conductance of presynaptic voltage-dependent calcium channels. After pre-treatment with magnesium, an increased speed of onset and a prolongation of the recovery period of neuromuscular blockade have been observed with other non-depolarizing neuromuscular blocking agent (NMBA) such as atracurium, vecuronium and rocuronium. Rocuronium is the currently preferred NMBA used as an alternative to succinylcholine for rapid tracheal intubation. As an alternative to succinylcholine, high doses of NMBA have been tested for rapid sequence intubation. This excessively high dose of rocuronium, however, prolongs the duration of the neuromuscular block and this may not be warranted in every surgical setting.

The reduction of onset time of rocuronium by magnesium pre-treatment can make intubation condition more rapid and much better clinically. It will thus be interesting to compare intubation conditions of a standard intubation dose of rocuronium after magnesium pre-treatment with high dose of rocuronium or standard dose of rocuronium.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing operation under general anesthesia
* American Society of Anesthesiologist physical status I or II
* 20-65 year old male or female

Exclusion Criteria:

* hepatic or renal dysfunction
* respiratory or cardiovascular dysfunction
* neurologic disorder
* neuromuscular disease
* pregnancy
* body mass index (BMI) >30 kg/m2 or <16.5 kg/m2
* anticipated difficult airway
* higher magnesium level than normal range in preoperative evaluation
* chronic medication with calcium channel blocker or magnesium
* history of known allergy to magnesium sulphate or any other study drugs

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
the intubating conditions | 1 minute during intervention
  The anesthesiologist also assessed the intubating conditions as per the intubation scoring system of the Good Clinical Research Practice guideline.

SECONDARY OUTCOMES:
mean arterial pressure (MAP) | 5 min before intubation, immediate before intubation, post-intubation 1, 2, 3, 4, and 5 min.
  They were recorded pre-induction (base line), just before intubation, and every minute thereafter for 5 min.
heart rate (HR) | 5 min before intubation, immediate before intubation, post-intubation 1, 2, 3, 4, and 5 min.
  They were recorded pre-induction (base line), just before intubation, and every minute thereafter for 5 min.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea